CLINICAL TRIAL: NCT02179801
Title: Screening Cardiovascular Patients for Aortic aNeurysms (SCAN)
Acronym: SCAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: I. Medizinischen Klinik und Poliklinik, Technical University of Munich (Unknown)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Hans-Henning Eckstein, Univ.-Prof. Dr. med. Hans-Henning Eckstein, Technical University of Munich
Other Study IDs: GES_SCAN
Record Dates: First submitted 2014-06-12; First posted 2014-07-02 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Abdominal Aortic Aneurysm; AAA
Keywords: Abdominal aortic aneurysm; AAA; Screening
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the cohort study SCAN (Screening Cardiovascular patients for Aortic aNeurysms) is to establish a screening programm for patients with a high risk for an AAA. Aortic aneurysms in these patients should be identified at an early stage and thereby AAA-associated mortality be decreased.

DETAILED DESCRIPTION:
A recently published meta-analysis showed a higher prevalence of aortic aneurysm (AAA) in men requiring treatment of coronary heart disaese compared to standard population. In women, however, the prevalence was not increased. Thus, the SCAN project addresses male patients who underwent coronary artery intervention in order to screen them for the presence of an AAA using duplex sonography.

The SCAN project involves the following elements:

1. Informing the patient with cardiovascular risk factors about the clinical picture of AAA
2. An ultrasound scan of the abdominal aorta in patients with an increased risk for AAA
3. Acquisition of patient data followed by a correlation analysis for the parameters presence of AAA and cardiovascular diseases

The cohort study is part of the SCAN project which is also conducted in an similar way by Catharina Ziekenhuis Eindhoven ClinicalTrials.gov Identifier:NCT01643317.

ELIGIBILITY:
Inclusion Criteria:

* men with coronary artery intervention (PTCA/stenting)
* at least 1 risk factor for AAA (hypertension, hyperlipidaemia, hyperuricemia, nicotine abuse,positive family history)

Exclusion Criteria:

* life expectancy less than 1 year
* inability to follow the instructions of the investigator (dementia, lack of time, insufficient understanding of the language)
* insufficient compliance

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men with coronary artery intervention (PTCA/stenting) and at least 1 risk factor for AAA (hypertension, hyperlipidaemia, hyperuricemia, nicotine abuse,positive family history.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of AAA | 1 year
  Ultrasound screen for the presence of an AAA

SECONDARY OUTCOMES:
Prevalence of AAA in the cohort requiring treatment | 1 year
  Measuring the AAA diameter
Correlation of risk factors for AAA with risk factors for coronary artery disease | 1 year
  Therefore the cardiovascular risk factors ( diabetes, hypertension, hyperlipidaemia, hyperuricemia, nicotine abuse, positive family history, obesity) will be requested.
Distribution of risk factors | 1 year
  Distribution of cardiovascular risk factors (diabetes, hypertension, hyperlipidaemia, hyperuricemia, nicotine abuse, positive family history, obesity) between patients with an without an AAA
Correlation of the number of treated vessels and AAA | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henning Eckstein, Univ.-Prof.Dr.med., Principal Investigator — Department for Vascular and Endovascular Surgery, Klinikum rechts der Isar der Technische Universität München; Karl-Ludwig Laugwitz, Univ.-Prof.Dr.med., Principal Investigator — I. Medizinischen Klinik und Poliklinik, Klinikum rechts der Isar der Technischen Universität München
Locations (2):
- Germany (2):
  - Klinikum rechts der Isar, Klinik und Poliklinik für Vaskuläre und Endovaskuläre Chirurgie, Munich, Bavaria
  - I. Medizinischen Klinik und Poliklinik, Klinikum rechts der Isar der Technischen Universität München, München, Bavaria